CLINICAL TRIAL: NCT05988385
Title: The Effects of Successful OSA Treatment on Memory and AD Biomarkers in Older Adults (ESSENTIAL) Study
Brief Title: The Effects of Successful OSA Treatment on Memory and AD Biomarkers in Older Adults Study
Acronym: ESSENTIAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); New York University (Other); University of Arizona (Other); University of Pittsburgh (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG080609
Record Dates: First submitted 2023-05-22; First posted 2023-08-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-06

CONDITIONS: Obstructive Sleep Apnea; Cognitive Decline
Keywords: Obstructive Sleep Apnea; OSA; Cognitive decline; Alzheimer Disease; AD; AD biomarkers; Positive Airway Pressure; PAP; CPAP; Oral appliance therapy; OAT; Positional therapy; Sleep-dependent memory
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Approximately 250 total patients (~63 per site) will be enrolled. In the 3-month wait-list control randomized trial, 200 patients will be randomized to one of two groups: i) a 3-month OSA treatment by any combination of PAP, OAT, and positional therapy that results in an "effective" AHI3a<15 (rapid multi-modal treatment RMMT); ii) a waitlist control group to receive treatment at the conclusion of the 3-month intervention period. The remaining 50, plus an additional ~50 (n~100 total) participants who declined treatment and were not interested in being randomized for the 3-month trial, or who have tried but failed treatment in the past, will serve as the "control" group for the 24-month follow-up period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 3-month OSA treatment (Active Comparator): A 3-month OSA treatment by any combination of PAP, OAT, and positional therapy that results in an "effective" AHI3a<15 (rapid multi-modal treatment RMMT).
  Interventions: Device: Positive airway pressure; Device: Oral appliance therapy; Device: Positional therapy
- Waitlist control group (Other): A waitlist control group to receive treatment at the conclusion of the 3-month intervention period.
  Interventions: Device: Positive airway pressure; Device: Oral appliance therapy; Device: Positional therapy

INTERVENTIONS:
Device: Positive airway pressure — Positive airway pressure (PAP) therapy is a sleep apnea treatment that uses a stream of compressed air to support the airway during sleep. With PAP therapy, a mask is worn during sleep and a portable machine gently blows pressurized room air from into your upper airway through a tube connected to the mask. This positive airflow helps keep the airway open, preventing the collapse that occurs during apnea, thus allowing normal breathing.
  Other Names: CPAP
Device: Oral appliance therapy — Oral appliance therapy involves the use of a dental appliance or oral mandibular advancement device that prevents the tongue from blocking the throat and/or advances the lower jaw forward. These devices help keep the airway open during sleep.
  Other Names: OAT; ProSomnus; Somnomed
Device: Positional therapy — A NightShift Sleep Positioner (Advanced Brain Monitoring) is a neck vibration device, FDA approved to treat positional sleep apnea. The device detects patient supine position and delivers a small vibratory signal to the back of the neck to prompt position change.
  Other Names: NightShift Sleep Positioner

SUMMARY:
The Effects of Successful OSA TreatmENT on Memory and AD BIomarkers in Older AduLts (ESSENTIAL) study is a 5-year, multicenter randomized open-label trial that will screen 400 cognitively normal older adults recruited from well-established sleep clinics at 4 academic medical centers, with newly diagnosed moderate-severe OSA. An expected 200 OSA patients will be then randomized to one of two groups: i) a 3-month OSA treatment by any combination of PAP, OAT, and positional therapy that results in an "effective" AHI4%< 10/hour and AHI3A<20/hour (see below); ii) a waitlist control group to receive treatment at the conclusion of the 3-month intervention period. Both groups will continue follow-up for 24 months on stable therapy to determine if sustained improvements in sleep are associated with improvement in cognitive function and AD biomarkers.

DETAILED DESCRIPTION:
The prevalence of Alzheimer disease (AD) is high and projected to increase. While there are multiple risk factors for AD, epidemiological data suggests that ~15% of AD risk may be attributed to sleep problems. Obstructive sleep apnea (OSA) is common among the elderly (30-55%), and the investigators have shown that cognitively normal older women with OSA have nearly double the risk of developing mild cognitive impairment (MCI) or dementia over 5 years. Further, the investigators have shown that in normal elderly, OSA predicts longitudinal increases in AD biomarkers. Our preliminary data also show that after positive airway pressure (PAP) withdrawal, OSA patients treated with PAP experienced significant overnight increases in plasma neurofilament light (NfL), a marker of neural injury. The present study is designed to overcome challenges identified in previous trials of treatment of OSA to slow cognitive decline and progression to AD. First, the most effective treatment for OSA, PAP therapy, has poor adherence (typically only 50% are adequately treated). Other common therapies include oral appliance therapy (OAT) which tends to be better tolerated but less effective. The investigators have piloted and propose for this study a rapid multimodal therapy initiation (RMMT) which ensures subjects will have effective therapy for their OSA that reduces OSA severity to AHI4%<10/hour and AHI3A (AKA pRDI) < 20/hour within 4 months. Second, most prior OSA treatment trials have focused primarily on symptomatic older adults (e.g. patients with MCI recruited from memory clinics), whereas early intervention in pre-symptomatic individuals may have stronger impact in preventing progression to AD. The investigators propose to enroll cognitively normal adults with newly diagnosed moderate-severe OSA (AHI4% >20/hour or AHI3A > 40/hour). Finally, selection of cognitive outcomes most responsive to OSA therapy has proved challenging. The Effects of Successful OSA TreatmENT on Memory and AD BIomarkers in Older AduLts (ESSENTIAL) study is a 5-year, multicenter randomized open-label trial that will screen 400 cognitively normal older adults (MoCA≥24, Clinical Dementia Rating [CDR]=0), ages 55-75, recruited from well-established sleep clinics at 4 academic medical centers, with newly diagnosed moderate-severe OSA (AHI4% >20/hour or AHI3A > 40/hour). An expected 200 OSA patients will be then randomized to one of two groups: i) a 3-month OSA treatment by any combination of PAP, OAT, and positional therapy that results in an "effective" AHI4%< 10/hour and AHI3A<20/hour (see below); ii) a waitlist control group to receive treatment at the conclusion of the 3-month intervention period. Both groups will continue follow-up for 24 months on stable therapy to determine if sustained improvements in sleep are associated with improvement in cognitive function and AD biomarkers. Both arms will include PSG and actigraphy, sleep-dependent memory and other cognitive evaluations, and blood draws at baseline, 3 and 24 months, with cognitive evaluation only at 12 months. Structural brain MRI will be performed at baseline. Because the investigators anticipate that 150 of 200 subjects will be well treated at 24 months, and 50 will not be, the investigators will additionally recruit ~50 subjects (on average 13 subjects per clinical site) with the same inclusion criteria who refuse treatment. These 50 subjects will perform baseline (blood draw and cognitive evaluations), 12-month (cognitive evaluation only), and 24-month (blood draw and cognitive evaluations) visits, allowing for a 24-month comparison of ~150 subjects with adequate treatment over 24 months to 100 subjects with inadequate treatment over 24 months. Our aims are: 1) To compare 3-month change in plasma AD biomarkers (NfL, p-tau, Aβ) in those randomized to OSA treatment and wait-list control groups (via both intention-to-treat and per-protocol analyses); 2) To test differences at 3 months in sleep-dependent declarative memory and cognitive scores (PACC and sub-domains) between the OSA treatment and wait-list control groups (via both intention-to-treat and per-protocol analyses); 3) To compare 24-month changes in AD biomarkers (NfL, p-tau, Aβ) and cognition in all successfully treated subjects and untreated controls.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively normal (TiCS ≥29)
* Age 55-85 years
* Moderate - severe OSA defined as AHI4 ≥20 events/hour or AHI3A>40/hr using a hypopnea criterion of a 4% oxygen desaturation (AHI4) or 3% oxygen desaturation and/or EEG arousal (AHI3A), or equivalent based on in-home testing - Testing must have been completed in past 12 months or confirmed by repeat test (EHR)
* Not currently on therapy for OSA and has not received treatment for OSA for at least 6months
* Able and willing to be treated for OSA (Treatment group)
* Fluency in English or Spanish

Exclusion Criteria:

* Documented diagnosis of chronic insomnia, or sleep onset insomnia based on Insomnia Severity Index - a answer of severe or very severe in the screening form
* Documented diagnosis of circadian rhythm disorder
* Any current use of supplemental oxygen
* Other sleep-related breathing disorders (central sleep apnea, etc) based on AASM criteria
* Current shift work involving night shift (regular work between 12am and 6am or night shift) within the past 6 mo
* Anticipated scheduled bariatric surgery within the next 3 months
* Chronic regular (> 2 nights per week) of cannabis for sleep
* Diagnosis of uncontrolled psychiatric disease in the last six months , and/or history of schizophrenia or bipolar disorder. Controlled conditions will include major depressive disorder, panic disorder, generalized anxiety disorder, OCD, substance use disorders, and alcohol abuse/dependence. (medical record/EHR). Personality disorders and neurodevelopmental disorders (e.g. autism, ADHD) are allowed if cognition is within normal limits.
* Taking methylphenidate for ADHD. Unless on stable dose which will be reviewed by the PI to determine.
* Taking GLP-1 agonist semaglutide (Ozempic, Wegovy, Rybelsus), or tirzepatide (Mounjaro, Zepbound), or similar for weightloss, and planning to lose an additional 20lbs or more at the time of enrollment. (Screening form/Electronic Medical Record) PI Discretion for determination of why they are taking the drug based on conversation with subject and medical chart, will be documented in form of Note-to-file in the subject's records
* Presence of other critical comorbid conditions that would lead to inability to complete the study protocol (including follow-up for 2 years), or that would affect cognition (e.g. clinically relevant endocrine or hematological conditions).
* Does not have a regular sleeping environment (i.e., sleeps in a different setting > 2 nights per week).
* Currently pregnant or planning to become pregnant.
* Prior diagnosis of a Central nervous system (CNS) disease, such as multiple sclerosis, stroke, Parkinson's disease, Alzheimer's disease, epilepsy, a loss of consciousness > 24 hours, or traumatic brain injury as identified by the Cumulative Illness Rating Scale for Geriatrics (CIRS). Participants who are diagnosed with MCI or Alzheimer's disease based on neuropsychological testing will be excluded. (CLINIC RECORDS/EHR). Delirium in the last 12 months.
* Near-miss or prior automobile accident "due to sleepiness" within the past 12 months.
* Employed as a commercial driver during the study (for example, bus drivers, train engineers, airplane pilots).
* Any use of neuroleptics, benzodiazepines, barbiturates, opiates or anti-amyloid therapies.
* Use of other cognitive enhancing drugs will also be excluded if initiated in the last 3 months, or not on stable dose.
* Consumption of >14 alcohol drinks per week, unless alcohol consumption can be reduced if initiated in the last 3 months

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in overnight memory retention on the A-B verbal paired associates task | 3 months
  Mean change in percent correct memory
Change in overnight memory retention on the A-B verbal paired associates task | 12 months
  Mean change in percent correct memory
Change in overnight memory retention on the A-B verbal paired associates task | 24 months
  Mean change in percent correct memory
Change in Aβ42/ Aβ40 ratio | 3 months
  Mean change in the Aβ42/ Aβ40 ratio in picograms per millimeter (pg/ml)
Change in Aβ42/ Aβ40 ratio | 24 months
  Mean change in the Aβ42/ Aβ40 ratio in picograms per millimeter (pg/ml)
Change in Plasma P-tau181 | 3 months
  Mean change in p-tau181 levels in the plasma in picograms per millimeter (pg/ml)
Change in Plasma P-tau181 | 24 months
  Mean change in p-tau181 levels in the plasma in picograms per millimeter (pg/ml)
Change in P-tau217 | 3 months
  Mean change in p-tau217 levels in the plasma in picograms per millimeter (pg/ml)
Change in P-tau217 | 24 months
  Mean change in p-tau217 levels in the plasma in picograms per millimeter (pg/ml)
Change in Neurofibrilary light (NfL) | 3 months
  Mean change in NfL levels in the plasma in picograms per millimeter (pg/ml)
Change in Neurofibrilary light (NfL) | 24 months
  Mean change in NfL levels in the plasma in picograms per millimeter (pg/ml)
Preclinical Cognitive Composite Score | 3 months
  Mean change in Preclinical Cognitive Composite Score.
Preclinical Cognitive Composite Score | 12 months
  Mean change in Preclinical Cognitive Composite Score.
Preclinical Cognitive Composite Score | 24 months
  Mean change in Preclinical Cognitive Composite Score.

SECONDARY OUTCOMES:
Change in Task-switching Accuracy | 3 months
  Change in Task-switching Mean Percent Accuracy
Change in Task-switching Accuracy | 12 months
  Change in Task-switching Mean Percent Accuracy
Change in Task-switching Accuracy | 24 months
  Change in Task-switching Mean Percent Accuracy
Change in Task-switching Reaction Time | 3 months
  Change in Task-switching Mean Reaction Time in milliseconds
Change in Task-switching Reaction Time | 12 months
  Change in Task-switching Mean Reaction Time in milliseconds
Change in Task-switching Reaction Time | 24 months
  Change in Task-switching Mean Reaction Time in milliseconds
Change in Psychomotor Vigilance Task (PVT) lapses | 3 months
  Mean change in number of lapses
Change in Psychomotor Vigilance Task (PVT) lapses | 12 months
  Mean change in number of lapses
Change in Psychomotor Vigilance Task (PVT) lapses | 24 months
  Mean change in number of lapses
Change in Psychomotor Vigilance Task (PVT) reaction time | 3 months
  Mean change in median reaction time in milliseconds.
Change in Psychomotor Vigilance Task (PVT) reaction time | 12 months
  Mean change in median reaction time in milliseconds.
Change in Psychomotor Vigilance Task (PVT) reaction time | 24 months
  Mean change in median reaction time in milliseconds.

OTHER OUTCOMES:
Cognitive Impairment Severity | Baseline
  Severity of cognitive impairment based on normed cutoffs with the National Alzheimer's Coordinating Centers Uniform Data Set-3 (UDS-3) assessment.
Cognitive Impairment Severity | 24 months
  Severity of cognitive impairment based on normed cutoffs with the National Alzheimer's Coordinating Centers Uniform Data Set-3 (UDS-3) assessment.
Clinical Dementia Rating (CDR) Scale (0-3) | Baseline
  Clinical Dementia Rating on a scale of 0-3 based on clinical assessment, 0 being no impairment, and 3 being severe impairment.
Sleepiness Score | Baseline
  Epworth Sleepiness Scale (ESS) Questionnaire Score. Higher scores mean more severe sleepiness.
Sleepiness Score | 3 months
  Epworth Sleepiness Scale (ESS) Questionnaire Score. Higher scores mean more severe sleepiness.
Sleepiness Score | 24 months
  Epworth Sleepiness Scale (ESS) Questionnaire Score. Higher scores mean more severe sleepiness.
Insomnia Severity | Baseline
  Insomnia Severity Index (ISI) Questionnaire Score. Higher scores mean more severe insomnia symptoms.
Insomnia Severity | 3 months
  Insomnia Severity Index (ISI) Questionnaire Score. Higher scores mean more severe insomnia symptoms.
Insomnia Severity | 24 months
  Insomnia Severity Index (ISI) Questionnaire Score. Higher scores mean more severe insomnia symptoms.
Psychiatric Symptom Questionnaires: Geriatric Depression Scale (GDS) | Baseline
  Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Psychiatric Symptom Questionnaires: Hamilton Anxiety Rating Scale (HAM-A) | Baseline
  Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Psychiatric Symptom Questionnaires: Clinician-Administered PTSD Scale (CAPS) | Baseline
  CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster: Criterion B (items 1-5); Criterion C (items 6-7); Criterion D (items 8-14); and, Criterion E (items 15-20). Severity scores range from 0-4, with 0 being absent to 4 being extreme/incapacitating.

CONTACTS AND LOCATIONS:
Overall Officials: Katie L Stone, PhD, Principal Investigator — California Pacific Medical Center Research Institute; Ricardo Osorio, MD, Principal Investigator — New York University; Andrew Varga, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - University of Arizona, Tucson, Arizona
  - New York University, New York, New York
  - Mount Sinai, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The final research data will be available in acceptable formats commonly accepted for documenting and supporting research findings. All data will be released and/or shared as soon as feasible without compromising privacy concerns, federal and state confidentiality concerns, proprietary interests, national security interests, or law enforcement activities. The final research data will not contain any patient identifiers. Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement.
Supporting Information: Study Protocol, ICF
Time Frame: Research data that documents, supports, and validates research findings will be available after the main findings from the final research data set are accepted for publication. We anticipate data will be available starting in January 2029 and will be available on an NIH-sponsored platform for as long as the agency supports it.
Access Criteria: Data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.